CLINICAL TRIAL: NCT01352481
Title: Early Intervention for Speech Sound Disorder in Very Preterm Children
Brief Title: Early Intervention in Very Preterm Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: RJ Baatenburg de Jong, MD, PhD, Head of Department, Erasmus Medical University Center, Department of Otorhinolatyngology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL33278.078.10
Record Dates: First submitted 2011-05-10; First posted 2011-05-12 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Prematurity; Speech Sound Disorder
Keywords: Speech sound development
MeSH Terms: conditions — Premature Birth; Speech Sound Disorder | interventions — Silver Sulfadiazine; Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Early parent-based speech intervention program
- Control group (No Intervention)
  Interventions: Other: Early parent-based speech intervention program

INTERVENTIONS:
Other: Early parent-based speech intervention program — Seven 1h sessions during a three-month period.
  Other Names: Prematurity, Speech Sound Disorder, Early Intervention

SUMMARY:
* The aim of the present study is to examine the effectiveness of a short, highly structured parent based speech intervention program on speech development in very preterm children with a Speech Sound Disorder (SSD) at 2 years of age.
* The hypothesis of this study is that early intervention on speech development is effective in improving the speech development in preterm children with SSD at 2 years of age compared to a no treatment group (usual care at this age).

ELIGIBILITY:
Inclusion Criteria:

* birth weight < 1500 grams or gestational age < 32 weeks
* singleton birth
* no major neurodevelopmental disabilities, and
* Dutch speaking family background

Ages: 24 Months to 27 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Number of acquired consonants produced by the child | 12 months after the onset of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical University Center, Rotterdam, Netherlands